CLINICAL TRIAL: NCT04471233
Title: Influence of Patient Sex on Pain Control and Multimodal Analgesia in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-0139
Record Dates: First submitted 2020-05-21; First posted 2020-07-15 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis; Pain, Postoperative
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Intervention is preoperative and 14 days postoperatively. Patients will be assigned to either multimodal analgesia regimen. No crossing over of patients will occur.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Care providers, and investigators will all be blinded to patient group identity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Multimodal analgesia regimen including pregabalin (Experimental): For the pregabalin group, patient will be provided with an oral preoperative pregabalin dose of 150mg on the day of surgery. Patient will continue pregabalin 75mg two times a day, for two weeks postoperatively. For both the intervention and control groups, the operative technique and additional perioperative analgesic modalities will follow a standard protocol
  Interventions: Other: Multimodal analgesia including pregabalin
- Multimodal analgesia regimen not including pregabalin (Active Comparator): For the non-pregabalin group, patient will be undergo total knee arthroplasty with the same operative technique and additional perioperative analgesic modalities will follow a standard protocol
  Interventions: Other: Multimodal analgesia not including pregabalin

INTERVENTIONS:
Other: Multimodal analgesia including pregabalin — Standardized protocol for our institution with multiple medications used for pain (NSAIDs, opioids, dexamethasone) and non-narcotic spinal. Patient will be provided with an preoperative pregabalin dose and will continue medication two weeks postoperatively.
  Arms: Multimodal analgesia regimen including pregabalin
Other: Multimodal analgesia not including pregabalin — Standardized protocol for our institution with multiple medications used for pain (NSAIDs, opioids, dexamethasone) and non-narcotic spinal.
  Arms: Multimodal analgesia regimen not including pregabalin

SUMMARY:
The purpose of this study is to examine the influence of sex on postoperative pain, following total knee arthroplasty (TKA). Patients will first be stratified by sex and then be randomized into one of two multimodal analgesic regimen (MAR), which differ in presence of pregabalin. We hypothesize that that acute postoperative pain scores are different over time between males and females and between multimodal analgesic regimens following TKA. Investigators will be blinded to which multimodal group patients are in. Patients will complete surveys in the office, during their hospital stay, and at followup intervals for up to six months.

DETAILED DESCRIPTION:
The overall goal of this study is to better understand the influence of patient-sex on postoperative pain perception in men versus women following total knee arthroplasty (TKA) utilizing two different multimodal analgesia regimens.

Pregabalin is a neuromuscular antagonist of voltage gated calcium channels at the post-synaptic dorsal horns in the spinal cord and brain. It binds to the alpha-2-delta subunit and interrupts pain signal transmission. The use of pregabalin as part of multimodal pain control has been associated with a decrease in postoperative opioid use.

This will be a randomized, single-blinded control trial in which patients either will or will not receive pregabalin as part of their multimodal analgesia regimen following TKA. It will be performed at a single institution, with multiple tertiary academic centers.

Patients will first be grouped according to their sex, then randomized into one of two arms:

1. Multimodal analgesia regimen including pregabalin;
2. Multimodal analgesia regimen not including pregabalin.

For the intervention group, patient will be provided with an oral preoperative pregabalin dose of 150mg on the day of surgery. Patient will continue pregabalin 75mg two times a day, for two weeks postoperatively. For both both groups, the operative technique and additional perioperative analgesic modalities will follow a standard protocol.

Primary Endpoint: Acute postoperative pain difference (up to 72 hours), measured by 100mm visual analogue scale (VAS) while at rest and mobilization, between males and females and between multimodal analgesic regimens in patients undergoing TKA.

Secondary Endpoints:

* Pain control measured by 100mm visual analogue scale (VAS) while at rest and mobilization.
* Pain control additionally measured by morphine equivalent units (MEq).
* Number of postoperative days to opioid cessation.
* Pain measured by Knee Injury and Osteoarthritis Outcome Score (KOOS).
* Physical function measured by KOOS, physical component summary (PCS-12) of VR-12.
* Mental health measured by mental component summary (MCS-12) of VR-12.
* Safety will be tracked by adverse reactions reported or observed by investigators. These will be collected via patient communication and review of the medical record.
* Additionally, severity of common short-term postoperative complications like nausea, vomiting, dizziness, and sedation will be assessed by 100mm VAS.

The study recruitment phase is estimated to last for 6 months. Subject followup is 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, age 18-80
4. Undergoing primary unilateral TKA for primary osteoarthritis
5. English speaking
6. Patients whose primary residence is in a home and not a facility or rehabilitation center.

Exclusion Criteria:

1. Chronic (>6 months) use of neuromodulators pregabalin or gabapentin.
2. Pregnancy or lactation
3. Prior history of adverse reactions to pregabalin
4. Coexisting chronic pain condition rated ≥50mm on 100-mm VAS requiring narcotics.
5. Coexisting condition leading to sedation or dizziness
6. Kidney disease
7. History of angioedema
8. History of depression with suicidal ideation.
9. Extensive history of opioid/ substance use and/or abuse.
10. Receiving active or maintenance treatment for cancer or solid organ and/or marrow transplant.
11. Patient staying less than one night in the hospital.
12. Patients with a history of chronic obstructive pulmonary disease (COPD) with supplementary oxygen requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility will be based on biological sex
Enrollment: 250 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Assess influence of sex and multimodal analgesia regimens on acute postoperative pain scores at 48 hours postoperatively, in patients undergoing TKA. | 48 hours
  Pain control measured by 100mm visual analogue scale (VAS) while at rest 48 hours after the procedure.

SECONDARY OUTCOMES:
Assess how sex differences and multimodal analgesia regimens influence physical function | 26 weeks
  -Pain measured by Knee Injury and Osteoarthritis Outcome Score (KOOS) of week 4, week 12, week 26 postoperatively, compared to baseline.
Assess how sex differences and multimodal analgesia regimens influence postoperative narcotic medication use | 72 hours
  Pain control additionally measured by morphine equivalent units (MEq) for 24, 48, and 72 hours after the end of the procedure.
Assess how sex differences and multimodal analgesia regimens influence postoperative narcotic medication cessation | 2 weeks
  -Number of postoperative days to opioid cessation.
Assess how sex differences and multimodal analgesia regimens influence chronic postoperative pain | 26 weeks
  -Chronic: Pain control measured by 100mm visual analogue scale (VAS) (0 corresponding to no pain and 100 corresponding to worst possible pain) while at rest and mobilization at week 1, week 2, week 4-6, week 12, week 26 postoperatively.
Assess how sex differences and multimodal analgesia regimens influence mental health | week 26
  -Mental health measured by mental component summary (MCS-12) of VR-12 of week 2, week 4, week 12, week 26 postoperatively, compared to baseline.
Assess how sex differences and multimodal analgesia regimens influence physical function | 26 weeks
  -Physical function measured physical component summary (PCS-12) of Veterans Rand-12 (VR-12) at week 2, week 4, week 12, week 26 postoperatively, compared to baseline.
Assess how sex differences and multimodal analgesia regimens influence range of motion (ROM) | 26 weeks
  Range of Motion (ROM) of week 2, week 4, week 12, week 26 postoperatively, compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Danoff, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health Orthopedic Institute at Great Neck, Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartley EJ, Fillingim RB. Sex differences in pain: a brief review of clinical and experimental findings. Br J Anaesth. 2013 Jul;111(1):52-8. doi: 10.1093/bja/aet127. PMID 23794645
- [Background] Berkley KJ. Sex differences in pain. Behav Brain Sci. 1997 Sep;20(3):371-80; discussion 435-513. doi: 10.1017/s0140525x97221485. PMID 10097000
- [Result] Anderson GD. Gender differences in pharmacological response. Int Rev Neurobiol. 2008;83:1-10. doi: 10.1016/S0074-7742(08)00001-9. PMID 18929073
- [Derived] Sodhi N, Qilleri A, Aprigliano C, Danoff JR. One Size Does Not Fit All: Women Experience More Pain Than Men After Total Knee Arthroplasty. J Arthroplasty. 2025 Apr;40(4):880-886. doi: 10.1016/j.arth.2024.09.028. Epub 2024 Sep 20. PMID 39307204